CLINICAL TRIAL: NCT01359319
Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Single and Repeat Doses of Sialic Acid Extended Release (SA-ER) Tables in Patients With Hereditary Inclusion Body Myopathy (HIBM)
Brief Title: Safety and Pharmacokinetics of Sialic Acid Tables in Patients With Hereditary Inclusion Body Myopathy (HIBM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX001-CL101
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-02

CONDITIONS: Hereditary Inclusion Body Myopathy (HIBM)
Keywords: Phase 1 Safety and Pharmacokinetic Study
MeSH Terms: conditions — Distal myopathy, Nonaka type | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 650 mg (single dose only) (Experimental): Each patient will be sequentially assigned to a specific dose level and will receive two single-dose exposures at that same dose level (fasted and fed). The low-dose cohorts will be filled before assigning higher-dose cohorts. The patient will then be assigned to receive one repeat-dose regimen. The lower-dose repeat-dose cohorts will be filled before proceeding to higher repeat-dose levels.
  Interventions: Drug: Sialic Acid Extended Release (SA-ER) Tablets
- 1,950 mg (single and repeat dose) (Experimental): Each patient will be sequentially assigned to a specific dose level and will receive two single-dose exposures at that same dose level (fasted and fed). The low-dose cohorts will be filled before assigning higher-dose cohorts. The patient will then be assigned to receive one repeat-dose regimen. The lower-dose repeat-dose cohorts will be filled before proceeding to higher repeat-dose levels.
  Interventions: Drug: Sialic Acid Extended Release (SA-ER) Tables
- 2,925 mg (single and repeat dose) (Experimental): Each patient will be sequentially assigned to a specific dose level and will receive two single-dose exposures at that same dose level (fasted and fed). The low-dose cohorts will be filled before assigning higher-dose cohorts. The patient will then be assigned to receive one repeat-dose regimen. The lower-dose repeat-dose cohorts will be filled before proceeding to higher repeat-dose levels.
  Interventions: Drug: Sialic Acid Extended Release (SA-ER) Tablets
- 4,875 mg (single and repeat dose) (Experimental): Each patient will be sequentially assigned to a specific dose level and will receive two single-dose exposures at that same dose level (fasted and fed). The low-dose cohorts will be filled before assigning higher-dose cohorts. The patient will then be assigned to receive one repeat-dose regimen. The lower-dose repeat-dose cohorts will be filled before proceeding to higher repeat-dose levels.
  Interventions: Drug: Sialic Acid Extended Release (SA-ER) Tablets
- 6,000 mg (single and repeat dose) (Experimental): Each patient will be sequentially assigned to a specific dose level and will receive two single-dose exposures at that same dose level (fasted and fed). The low-dose cohorts will be filled before assigning higher-dose cohorts. The patient will then be assigned to receive one repeat-dose regimen. The lower-dose repeat-dose cohorts will be filled before proceeding to higher repeat-dose levels.
  Interventions: Drug: Sialic Acid Extended Release (SA-ER) Tablets

INTERVENTIONS:
Drug: Sialic Acid Extended Release (SA-ER) Tablets — Patients will receive SA-ER tablets orally at one of five (5) dose levels in the single-dose phase,phase and one of four (4) dose levels in the repeat-dose phase. During repeat dosing, the total daily dose will be divided evenly into three doses given in the morning, in the evening, and at bedtime (qHS). No placebo or active comparator will be administered and the study drug will be administered on an open-label basis.
  Arms: 650 mg (single dose only)
Drug: Sialic Acid Extended Release (SA-ER) Tables — PPatients will receive SA-ER tablets orally at one of five (5) dose levels in the single-dose phase,phase and one of four (4) dose levels in the repeat-dose phase. During repeat dosing, the total daily dose will be divided evenly into three doses given in the morning, in the evening, and at bedtime (qHS). No placebo or active comparator will be administered and the study drug will be administered on an open-label basis.
  Arms: 1,950 mg (single and repeat dose)
Drug: Sialic Acid Extended Release (SA-ER) Tablets — Patients will receive SA-ER tablets orally at one of five (5) dose levels in the single-dose phase,phase and one of four (4) dose levels in the repeat-dose phase. During repeat dosing, the total daily dose will be divided evenly into three doses given in the morning, in the evening, and at bedtime (qHS). No placebo or active comparator will be administered and the study drug will be administered on an open-label basis.
  Arms: 2,925 mg (single and repeat dose)
Drug: Sialic Acid Extended Release (SA-ER) Tablets — Patients will receive SA-ER tablets orally at one of five (5) dose levels in the single-dose phase,phase and one of four (4) dose levels in the repeat-dose phase. During repeat dosing, the total daily dose will be divided evenly into three doses given in the morning, in the evening, and at bedtime (qHS). No placebo or active comparator will be administered and the study drug will be administered on an open-label basis.
  Arms: 4,875 mg (single and repeat dose)
Drug: Sialic Acid Extended Release (SA-ER) Tablets — Patients will receive SA-ER tablets orally at one of five (5) dose levels in the single-dose phase,phase and one of four (4) dose levels in the repeat-dose phase. During repeat dosing, the total daily dose will be divided evenly into three doses given in the morning, in the evening, and at bedtime (qHS). No placebo or active comparator will be administered and the study drug will be administered on an open-label basis.
  Arms: 6,000 mg (single and repeat dose)

SUMMARY:
Hereditary Inclusion Body Myopathy (HIBM) is a severe progressive metabolic myopathy caused by a defect in the biosynthetic pathway for sialic acid (SA), a critical component of many muscle proteins, resulting in a deficiency in SA in the muscles of HIBM patients.

The effective replacement of the missing SA substrate is theoretically simple, and, in animal models, replacement with SA showed significant restoration of sialylation biochemistry and excellent reduction in muscle disease. These data show that replacement can achieve significant clinical benefit in muscle pathology, function, and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years to 70 years of age.
2. Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
3. Must have a documented diagnosis, confirmed by genetic testing, of hereditary inclusion body myopathy (HIBM), also known as distal myopathy, rimmed vacuoles (DMRV), or Nonaka myopathy due to demonstrated mutations in gene encoding the GNE/MNK enzyme.
4. Willing and able to comply with all study procedures, including multiple overnight stays at a hospital unit or Phase 1 unit.
5. Sexually active subjects must be willing to use an acceptable method of contraception (i.e double barrier method)while participating in the study and for 30 days after receiving the last dose of SA-ER.
6. Females of childbearing potential must have a negative pregnancy test at screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had bilateral tubal ligation at least 1 year prior to screening, or who have had total hysterectomy.

Exclusion Criteria:

1. Pregnant or breastfeeding at screening or planning to become pregnant (self or partner) at any time during the study.
2. Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
3. Ingestion of ManNAc, sialic acid, or related metabolites or sialic acid donors that provide this substrate in either chemical or nutritional supplement form during the 30 days prior to screening. If ManNAc or other substrate was used more than 30 days prior to screening, the time period of use, the compound used, and the dose and dose regimen should be recorded in the patient's history. If a patient has been on substrate replacement therapy in the past, the investigator must consider the potential confounding effects of this therapy before enrolling the patient.
4. Presence of a condition the severity and acuity of which, in the opinion of the investigator, warrant immediate surgical intervention or other treatment.
5. Presence or history of any hypersensitivity to SA or its excipients that, in the judgment of the investigator, places the subject at increased risk for adverse effects.
6. Presence of a concurrent disease or condition that would interfere with study participation or affect safety such as swallowing difficulties.
7. Presence or history of any condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study.
8. Serum transaminase (ALT, AST, GGT) levels > 3 x upper limit of normal (ULN) or serum creatinine > 2.0 mg/dL.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of repeated doses of Sialic Acid - Extended Release (SA-ER) tablets in patients with HIBM | Each patient may participate approximately 4-6 weeks total, including 2 single dose (fast/fed) treatment periods followed by a 7-day repeat treatment period.
  Safety will be evaluated in terms of the incidence and frequency of treatment-emergent adverse events (TEAEs), including clinically significant changes from baseline to scheduled timepoints in clinical laboratory values, vital signs, or physical and neurologic examination findings. Medical history and reported clinical symptoms, including increasing muscle weakness, fatigue, or pain.

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of SA-ER after single and repeated dosing. | Multiple pharmacokinetic (serum) samples will be taken during the study, at baseline, after each single dose administration, and at the final day of the 7 day repeat dose period.
  Evaluation of the pharmacokinetics of SA-ER will include Cmax, the AUC of single doses, and steady-state levels of free, soluble sialic acid in serum after repeated dosing.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - West Coast Clinical Trials, Costa Mesa, California
  - Clinilabs, New York, New York